CLINICAL TRIAL: NCT00190333
Title: Evaluation of the Therapeutic Effects of Escitalopram in Pulmonary Hypertension, Either Primary or Associated
Brief Title: Serotonin Transporter Inhibitor Escitalopram in Pulmonary Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Isabelle BRINDEL, Department of Clinical Research of developpement
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P020305
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2007-03

CONDITIONS: Pulmonary Hypertension
Keywords: pulmonary hypertension; 6 minutes walking test; serotonin; primary or associated pulmonary hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Active Comparator)
  Interventions: Drug: escitalopram

INTERVENTIONS:
Drug: escitalopram — escitalopram

SUMMARY:
This is a Phase III, multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy of escitalopram (30 mg/day) in two parallel groups (randomization ratio, escitalopram 2/placebo 1).

DETAILED DESCRIPTION:
Primary objective: to evaluate the efficacy of oral escitalopram at the dosage of 30 mg/day for 16 weeks on the 6-minute walking test in patients with pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all the criteria listed below will be considered for study inclusion:

* Male or female older than 18 years of age
* Meeting World Health Organization (WHO) criteria for pulmonary hypertension (mean pulmonary arterial pressure [PAP] > 25 mmHg at rest and pulmonary capillary wedge pressure < 15 mmHg during right heart catheterization):

  * primary pulmonary hypertension (sporadic or familial), or
  * pulmonary hypertension associated with connective tissue diseases, or
  * pulmonary hypertension associated with HIV infection, or
  * pulmonary hypertension associated with use of appetite suppressants or other toxic compounds, or
  * pulmonary hypertension associated with shunting through a congenital heart defect surgically treated
* Class II or III in the NYHA classification scheme
* With a 6-minute walking test distance between 40% and 80% of theoretical values (approximately 50 and 480 m)
* On conventional treatment, with no change in this treatment during the last month preceding the study. Conventional treatment includes calcium antagonists or beraprost.
* Subject who consents to participate in the study.

Exclusion Criteria:

Subjects with any of the following clinical features will not be included in the study:

* Pulmonary hypertension related to aortic or mitral valve disease, or extrinsic pulmonary vein compression
* Pulmonary hypertension related to hypoxia from respiratory disease with a total lung capacity < 70% or Tiffeneau index < 60% upon testing within the last 6 months (chronic obstructive lung disease, interstitial disease, sleep apnea syndrome, alveolar hypoventilation, chronic exposure to high altitudes, neonatal lung disease, or alveolar capillary dysplasia)
* Pulmonary hypertension associated with portal hypertension
* Pulmonary hypertension secondary to chronic thrombosis and/or embolism (occlusion of the proximal or distal pulmonary arteries by thrombosis)
* In the 6-minute walking test, inability to walk for 6 minutes, for any reason, or walking distance of less than 50 m
* Pregnancy, lactation, women of childbearing potential (if needed, effective contraception will be prescribed)
* History of hypersensitivity to citalopram or to medications structurally related to citalopram
* Treatment with another investigational drug within the 3 months preceding study inclusion
* Cardiovascular, hepatic, neurological or endocrine disease that is clinically significant, or any other significant disease that may interfere with the study protocol or with the interpretation of study findings
* History of drug or alcohol abuse
* Liver failure (except abnormalities related to the right ventricular failure)
* Kidney failure
* Mental status preventing the patient from understanding the nature, objectives, and possible consequences of the study
* Non stabilized psychiatric disorders
* Subject unable to comply with protocol-related constraints (e.g., uncooperative, unable to attend follow-up visits, and probably unable to complete the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of oral escitalopram at the dosage of 30 mg/day on the 6-minute walking test in patients with pulmonary hypertension | for 16 weeks

SECONDARY OUTCOMES:
To evaluate the efficacy of escitalopram in improving hemodynamic parameters (right heart catheterization; decision of doing right heart catheterization belonging to the investigators) | after 16 weeks
To evaluate the efficacy of escitalopram in improving the New York Heart Association (NYHA) class | after 16 weeks
To evaluate the efficacy of escitalopram in improving the dyspnea (visual analog scale) | after 16 weeks
To evaluate the efficacy of escitalopram in improving the quality of life | after 16 weeks
To evaluate the efficacy of escitalopram in reducing exacerbations of signs or symptoms of the disease that would otherwise require hospital admission or treatment intensification, particularly treatment with bosentan or IV administration of epoprostenol | after 16 weeks
To evaluate the safety of escitalopram, alone or on top of associated drugs | after 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gerald SIMONNEAU, MD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (9):
- France (9):
  - Louis Pradel Hospital, Bron
  - Antoine Beclere Hospital, Clamart
  - Henri Mondor Hospital, Créteil
  - Michallon Hospital, Grenoble
  - Sainte Marguerite Hospital, Marseille
  - Haut Lévèque Hospital, Pessac
  - Hautepierre Hospital, Strasbourg
  - Rangueil Hospital, Toulouse
  - Brabois Hospital, Vandœuvre-lès-Nancy